CLINICAL TRIAL: NCT01368042
Title: Quality of Life in Greek Hemodialysis Patients Receiving Zemplar i.v (QualitiZe)
Brief Title: Quality of Life in Greek Hemodialysis Patients Receiving Zemplar Intravenous
Acronym: QUALITIZE
Status: Completed | Type: Observational
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Other Study IDs: P12-776
Record Dates: First submitted 2011-06-06; First posted 2011-06-07 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Kidney Disease; Secondary Hyperparathyroidism
Keywords: Quality of Life changes; Secondary Hyperparathyroidism; Chronic Kidney Disease; Hemodialysis; Paricalcitol intravenous treatment
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperparathyroidism, Secondary

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Kidney Disease, Secondary Hyperpathyroidism: All eligible participants treated with paricalcitol iv according to the approved Summary of Product Characteristics (SmPC)

SUMMARY:
The purpose of this study is to assess health-related Quality of Life (QoL) changes in participants with chronic kidney disease (CKD) and secondary hyperparathyroidism (sHPT) undergoing hemodialysis and receiving paricalcitol intravenous (iv).

DETAILED DESCRIPTION:
The scientific purpose of this study is to obtain data on the use of paricalcitol iv in real-life clinical practice and the effect it has on participant health-related QoL. In this study, paricalcitol iv will be prescribed on an on-label basis in an everyday setting. The RAND 36-Item Health Survey results will be collected for a 6-month period (every 3 months) in order to assess the effect of paricalcitol iv on participant health-related QoL.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic kidney disease stage 5 undergoing hemodialysis and receiving paricalcitol iv for more than 1 month.
2. Patients with a RAND 36-Item Health Survey completed 10 to 35 days before paricalcitol iv initiation
3. Patients with baseline parathormone ≥ 300 pg/mL
4. Patients willing to give their informed consent to participate in the study.
5. Patients should not receive vitamin D-related compounds or cinacalcet for 3 months prior to entering the study
6. Patients must be on steady regimen for anemia, hypertension and diabetes for the past 30 days

Exclusion Criteria:

1. Patients with a history of clinically significant intolerance or sensitivity to vitamin D or any ingredients of the product.
2. Patients with persistent hypercalcemia or evidence of vitamin D toxicity.
3. Patients with a continuous increase in serum (calcium x phosphorus) product greater than 65.
4. Pregnant or lactating female patients.
5. Patients who have previously undergone parathyroidectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease stage 5 on hemodialysis and diagnosed with secondary hyperparathyroidism, who were prescribed paricalcitol intravenous according to the approved Summary of Product Characteristics
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2011-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos Argyropoulos, MD, Study Chair — AbbVie
Locations (11):
- Greece (11):
  - Site Reference ID/Investigator# 56803, Arta
  - Site Reference ID/Investigator# 53424, Athens
  - Site Reference ID/Investigator# 53425, Larissa
  - Site Reference ID/Investigator# 56805, Lefkada
  - Site Reference ID/Investigator# 56802, Melíssia
  - Site Reference ID/Investigator# 66291, Pátrai
  - Site Reference ID/Investigator# 56809, Pátrai
  - Site Reference ID/Investigator# 50442, Pylaia Thessaloniki
  - Site Reference ID/Investigator# 77554, Thessaloniki
  - Site Reference ID/Investigator# 77553, Thessaloniki
  - Site Reference ID/Investigator# 53422, Volos

REFERENCES:
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 265 participants enrolled, 11 participants were considered to have protocol deviations and were excluded from the enrolled population and from all study-related analyses. A total of 254 participants were included in all of the study analyses.
Period: Overall Study
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Started | 265
Completed | 235
Not Completed | 30
Not completed — Death | 14
Not completed — Protocol Violation | 11
Not completed — Lost to Follow-up | 4
Not completed — Transplanted | 1

BASELINE CHARACTERISTICS:
Population: All participants in the enrolled population, regardless of whether or not they completed the study (i.e., the 6-month post-enrollment follow-up). Of the 265 participants enrolled, 11 were considered to have protocol deviations and were excluded from the enrolled population; therefore, 254 participants were included in the study analyses.
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95
  Male | 159

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 6 Months Post-enrollment in RAND 36-Item Health Survey 'Physical Functioning' Scale Scores
Description: The RAND 36-Item Health Survey questionnaire is self-completed by the participant and includes 36 questions that assess 8 different scales, including physical functioning. The scores for each scale range from 0 to 100, with 0 representing the worst possible state of physical functioning and 100 representing the best possible state of physical functioning. Baseline was 10 to 35 days prior to starting treatment with paricalcitol iv; enrollment was at least 1 month after starting treatment with paricalcitol iv. The change from baseline to the 6-month post-enrollment visit was calculated as the 6-month post-enrollment visit score minus the baseline score.
Time Frame: Baseline, 6 months post-enrollment
Population: All participants in the enrolled population with an available RAND 36-Item Health Survey score at the study timepoints. Of the 265 participants enrolled, 11 were considered to have protocol deviations and were excluded from the enrolled population; therefore, 254 participants were included in the study analyses.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
scores on a scale
  Baseline (n=253) | 49.3 (30.0)
  6 months post-enrollment (n=235) | 56.2 (30.4)
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p = 0.03, Wilcoxon signed rank test-paired samples; Mean Difference (Final Values) = 5.7, Standard Deviation 32.9 — n=234 (paired samples)

2. Primary Outcome: Change From Baseline to 6 Months Post-enrollment in RAND 36-Item Health Survey 'Role Limitations Due to Physical Health' Scale Scores
Description: The RAND 36-Item Health Survey questionnaire is self-completed by the participant and includes 36 questions that assess 8 different scales, including role limitations due to physical health. The scores for each scale range from 0 to 100, with 0 representing the worst possible score and 100 representing the best possible score. Baseline was 10 to 35 days prior to starting treatment with paricalcitol iv; enrollment was at least 1 month after starting treatment with paricalcitol iv. The change from baseline to the 6-month post-enrollment visit was calculated as the 6-month post-enrollment visit score minus the baseline score.
Time Frame: Baseline, 6 months post-enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
scores on a scale
  Baseline (n=253) | 41.5 (43.2)
  6 months post-enrollment (n=232) | 49.9 (46.4)
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p = 0.05, Wilcoxon signed rank test-paired samples; Mean Difference (Final Values) = 7.3, Standard Deviation 57.2 — n=231 (paired samples)

3. Primary Outcome: Change From Baseline to 6 Months Post-enrollment in RAND 36-Item Health Survey 'Role Limitations Due to Emotional Problems' Scale Scores
Description: The RAND 36-Item Health Survey questionnaire is self-completed by the participant and includes 36 questions that assess 8 different scales, including role limitations due to emotional problems. The scores for each scale range from 0 to 100, with 0 representing the worst possible score and 100 representing the best possible score. Baseline was 10 to 35 days prior to starting treatment with paricalcitol iv; enrollment was at least 1 month after starting treatment with paricalcitol iv. The change from baseline to the 6-month post-enrollment visit was calculated as the 6-month post-enrollment visit score minus the baseline score.
Time Frame: Baseline, 6 months post-enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
scores on a scale
  Baseline (n=253) | 43.5 (44.4)
  6 months post-enrollment (n=232) | 54.2 (46.0)
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p = 0.003, Wilcoxon signed rank test-paired samples; Mean Difference (Final Values) = 10.8, Standard Deviation 56.4 — n=231 (paired samples)

4. Primary Outcome: Change From Baseline to 6 Months Post-enrollment in RAND 36-Item Health Survey 'Energy/Fatigue' Scale Scores
Description: The RAND 36-Item Health Survey questionnaire is self-completed by the participant and includes 36 questions that assess 8 different scales, including energy/fatigue. The scores for each scale range from 0 to 100, with 0 representing the worst possible score and 100 representing the best possible score. Baseline was 10 to 35 days prior to starting treatment with paricalcitol iv; enrollment was at least 1 month after starting treatment with paricalcitol iv. The change from baseline to the 6-month post-enrollment visit was calculated as the 6-month post-enrollment visit score minus the baseline score.
Time Frame: Baseline, 6 months post-enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
scores on a scale
  Baseline (n=254) | 50.2 (24.8)
  6 months post-enrollment (n=235) | 63.8 (23.6)
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test-paired samples; Mean Difference (Final Values) = 12.5, Standard Deviation 30.5 — n=235 (paired samples)

5. Primary Outcome: Change From Baseline to 6 Months Post-enrollment in RAND 36-Item Health Survey 'Emotional Well-Being' Scale Scores
Description: The RAND 36-Item Health Survey questionnaire is self-completed by the participant and includes 36 questions that assess 8 different scales, including emotional well-being. The scores for each scale range from 0 to 100, with 0 representing the worst possible score and 100 representing the best possible score. Baseline was 10 to 35 days prior to starting treatment with paricalcitol iv; enrollment was at least 1 month after starting treatment with paricalcitol iv. The change from baseline to the 6-month post-enrollment visit was calculated as the 6-month post-enrollment visit score minus the baseline score.
Time Frame: Baseline, 6 months post-enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
scores on a scale
  Baseline (n=254) | 59.4 (22.0)
  6 months post-enrollment (n=235) | 68.3 (22.6)
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test-paired samples; Mean Difference (Final Values) = 8.4, Standard Deviation 27.2 — n=235 (paired samples)

6. Primary Outcome: Change From Baseline to 6 Months Post-enrollment in RAND 36-Item Health Survey 'Social Functioning' Scale Scores
Description: The RAND 36-Item Health Survey questionnaire is self-completed by the participant and includes 36 questions that assess 8 different scales, including social functioning. The scores for each scale range from 0 to 100, with 0 representing the worst possible score and 100 representing the best possible score. Baseline was 10 to 35 days prior to starting treatment with paricalcitol iv; enrollment was at least 1 month after starting treatment with paricalcitol iv. The change from baseline to the 6-month post-enrollment visit was calculated as the 6-month post-enrollment visit score minus the baseline score.
Time Frame: Baseline, 6 months post-enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
scores on a scale
  Baseline (n=254) | 55.9 (28.6)
  6 months post-enrollment (n=235) | 67.2 (28.1)
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test-paired samples; Mean Difference (Final Values) = 10.3, Standard Deviation 35.3 — n=235 (paired samples)

7. Primary Outcome: Change From Baseline to 6 Months Post-enrollment in RAND 36-Item Health Survey 'Bodily Pain' Scale Scores
Description: The RAND 36-Item Health Survey questionnaire is self-completed by the participant and includes 36 questions that assess 8 different scales, including bodily pain. The scores for each scale range from 0 to 100, with 0 representing the worst possible score and 100 representing the best possible score. Baseline was 10 to 35 days prior to starting treatment with paricalcitol iv; enrollment was at least 1 month after starting treatment with paricalcitol iv. The change from baseline to the 6-month post-enrollment visit was calculated as the 6-month post-enrollment visit score minus the baseline score.
Time Frame: Baseline, 6 months post-enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
scores on a scale
  Baseline (n=253) | 57.1 (28.9)
  6 months post-enrollment (n=235) | 68.5 (28.5)
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test-paired samples; Mean Difference (Final Values) = 10.7, Standard Deviation 34.8 — n=234 (paired samples)

8. Primary Outcome: Change From Baseline to 6 Months Post-enrollment in RAND 36-Item Health Survey 'General Health Perceptions' Scale Scores
Description: The RAND 36-Item Health Survey questionnaire is self-completed by the participant and includes 36 questions that assess 8 different scales, including general health perceptions. The scores for each scale range from 0 to 100, with 0 representing the worst possible score and 100 representing the best possible score. Baseline was 10 to 35 days prior to starting treatment with paricalcitol iv; enrollment was at least 1 month after starting treatment with paricalcitol iv. The change from baseline to the 6-month post-enrollment visit was calculated as the 6-month post-enrollment visit score minus the baseline score.
Time Frame: Baseline, 6 months post-enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
scores on a scale
  Baseline (n=254) | 38.9 (17.8)
  6 months post-enrollment (n=235) | 39.5 (17.2)
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p = 0.38, Wilcoxon signed rank test-paired samples; Mean Difference (Final Values) = 0.3, Standard Deviation 20.9 — n=235 (paired samples)

9. Primary Outcome: Change From Baseline to 6 Months Post-enrollment in RAND 36-Item Health Survey 'Health Change' Item Scores
Description: The RAND 36-Item Health Survey questionnaire is self-completed by the participant and includes a single question pertaining to the participant's health change over the last year. The scores range from 0 to 100, with 100: much better than 1 year ago; 75: somewhat better than 1 year ago; 50: about the same; 25: somewhat worse than 1 year ago; 0: much worse than 1 year ago. Baseline was 10 to 35 days prior to starting treatment with paricalcitol iv; enrollment was at least 1 month after starting treatment with paricalcitol iv. The change from baseline to the 6-month post-enrollment visit was calculated as the 6-month post-enrollment visit score minus the baseline score.
Time Frame: Baseline, 6 months post-enrollment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
scores on a scale
  Baseline (n=254) | 50.6 (26.0)
  6 months post-enrollment (n=235) | 65.0 (27.1)
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p < 0.001, Wilcoxon signed rank test-paired samples; Mean Difference (Final Values) = 14.0, Standard Deviation 32.0 — n=235 (paired samples)

10. Primary Outcome: Change Per Month From Baseline to 6 Months Post-enrollment on the 8 Scales of the RAND 36-Item Health Survey
Description: The RAND 36-Item Health Survey questionnaire is self-completed by the participant and includes 36 questions that assess 8 different scales (physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, bodily pain, general health perception, health change). Baseline was 10 to 35 days prior to starting treatment with paricalcitol iv; enrollment was at least 1 month after starting treatment with paricalcitol iv. The change from baseline to the enrollment and post-enrollment visits was calculated as the visit score minus the baseline score. Linear models based on Generalized Estimating Equations (GEE) were used to assess the effect of time on change from baseline through enrollment, 3 months post-enrollment, and 6 months post-enrollment.
Time Frame: Baseline, enrollment, 3 months post-enrollment, 6 months post-enrollment
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: scores on a scale/month
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
scores on a scale/month
  Physical Functioning Scale | 0.67 [0.08 to 1.26]
  Role Functioning due to Physical Health Scale | 1.31 [0.24 to 2.38]
  Role Functioning due to Emotional Problems Scale | 1.42 [0.31 to 2.53]
  Energy/Fatigue Scale | 1.34 [0.82 to 1.87]
  Emotional well-being | 0.71 [0.26 to 1.16]
  Social Functioning Scale | 1.01 [0.36 to 1.66]
  Bodily Pain Scale | 1.69 [1.03 to 2.34]
  General Health Perceptions Scale | 0.11 [-0.27 to 0.50]
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Physical functioning scale; Test type: Superiority or Other; p = 0.03, Generalized Estimating Equation approach; Generalized Estimating Equation approach (autoregressive structure)
Statistical Analysis 2: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Role functioning due to physical health scale; Test type: Superiority or Other; p = 0.02, Generalized Estimating Equation approach; Generalized Estimating Equation approach (autoregressive structure)
Statistical Analysis 3: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Role functioning due to emotional problems scale; Test type: Superiority or Other; p = 0.01, Generalized Estimating Equation approach; Generalized Estimating Equation approach (autoregressive structure)
Statistical Analysis 4: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Energy/fatigue scale; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equation approach; Generalized Estimating Equation approach (autoregressive structure)
Statistical Analysis 5: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Emotional well-being scale; Test type: Superiority or Other; p = 0.002, Generalized Estimating Equation approach; Generalized Estimating Equation approach (autoregressive structure)
Statistical Analysis 6: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Social functioning scale; Test type: Superiority or Other; p = 0.002, Generalized Estimating Equation approach; Generalized Estimating Equation approach (autoregressive structure)
Statistical Analysis 7: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Bodily pain scale; Test type: Superiority or Other; p < 0.001, Generalized Estimating Equation approach; Generalized Estimating Equation approach (autoregressive structure)
Statistical Analysis 8: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; General health perceptions scale; Test type: Superiority or Other; p = 0.56, Generalized Estimating Equation approach; Generalized Estimating Equation approach (autoregressive structure)

11. Secondary Outcome: Change From Enrollment to 6 Months Post-enrollment in Urea Levels (mg/dL)
Description: Urea levels were recorded at each study visit prior to hemodialysis according to routine clinical practice and at the discretion of the physician. The change from enrollment (at least 1 month after starting treatment with paricalcitol iv) to the 6-month post-enrollment visit was calculated as the 6-month post-enrollment visit value minus the enrollment value.
Time Frame: Enrollment, 6 months post-enrollment
Population: All participants in the enrolled population with available data at the study timepoints, regardless of whether or not they completed the study (i.e., the 6-month post-enrollment follow-up). Of the 265 participants enrolled, 11 were considered to have protocol deviations and excluded; therefore, 254 participants were included in the study analyses.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
mg/dL
  Enrollment (n=254) | 147.7 (42.3)
  6 month post-enrollment (n=235) | 139.9 (43.1)
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p = 0.001, Wilcoxon signed rank test-paired samples; Mean Difference (Final Values) = -9.0, Standard Deviation 41.6 — n=235 (paired samples)

12. Secondary Outcome: Change From Enrollment to 6 Months Post-enrollment in Creatinine Levels (mg/dL)
Description: Creatinine levels were recorded at each study visit prior to hemodialysis according to routine clinical practice and at the discretion of the physician. The change from enrollment (at least 1 month after starting treatment with paricalcitol iv) to the 6-month post-enrollment visit was calculated as the 6-month post-enrollment visit value minus the enrollment value.
Time Frame: Enrollment, 6 months post-enrollment
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
mg/dL
  Enrollment (n=254) | 8.0 (2.7)
  6 months post-enrollment (n=235) | 8.3 (2.8)
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p = 0.03, Wilcoxon signed rank test-paired samples; Mean Difference (Final Values) = 0.2, Standard Deviation 1.4 — n=235 (paired samples)

13. Secondary Outcome: Change From Enrollment to 6 Months Post-enrollment in Calcium Levels (mg/dL)
Description: Calcium levels were recorded at each study visit prior to hemodialysis according to routine clinical practice and at the discretion of the physician. The change from enrollment (at least 1 month after starting treatment with paricalcitol iv) to the 6-month post-enrollment visit was calculated as the 6-month post-enrollment visit value minus the enrollment value.
Time Frame: Enrollment, 6 months post-enrollment
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
mg/dL
  Enrollment (n=254) | 9.0 (0.8)
  6 months post-enrollment (n=235) | 9.1 (0.9)
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p = 0.06, Wilcoxon signed rank test-paired samples; Mean Difference (Final Values) = 0.1, Standard Deviation 0.9 — n=235 (paired samples)

14. Secondary Outcome: Change From Enrollment to 6 Months Post-enrollment in Phosphorous Levels (mg/dL)
Description: Phosphorous levels were recorded at each study visit prior to hemodialysis according to routine clinical practice and at the discretion of the physician. The change from enrollment (at least 1 month after starting treatment with paricalcitol iv) to the 6-month post-enrollment visit was calculated as the 6-month post-enrollment visit value minus the enrollment value.
Time Frame: Enrollment, 6 months post-enrollment
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
mg/dL
  Enrollment (n=254) | 5.2 (1.4)
  6 months post-enrollment (n=234) | 5.2 (1.5)
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p = 0.84, Wilcoxon signed rank test-paired samples; Mean Difference (Final Values) = -0.06, Standard Deviation 1.7 — n=234 (paired samples)

15. Secondary Outcome: Change From Enrollment to 6 Months Post-enrollment in Calcium-Phosphorous (Ca×P) Product Levels (mg˄2/dL˄2)
Description: Ca×P product levels were recorded at each study visit prior to hemodialysis according to routine clinical practice and at the discretion of the physician. The change from enrollment (at least 1 month after starting treatment with paricalcitol iv) to the 6-month post-enrollment visit was calculated as the 6-month post-enrollment visit value minus the enrollment value.
Time Frame: Enrollment, 6 months post-enrollment
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mg˄2/dL˄2
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
mg˄2/dL˄2
  Enrollment (n=254) | 46.6 (14.4)
  6 months post-enrollment (n=234) | 47.1 (14.8)
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p = 0.67, Wilcoxon signed rank test-paired samples; Mean Difference (Final Values) = -0.01, Standard Deviation 16.5 — n=234 (paired samples)

16. Secondary Outcome: Change From Enrollment to 6 Months in Parathyroid Hormone (PTH) Levels (pg/mL)
Description: PTH levels were recorded at each study visit prior to hemodialysis according to routine clinical practice and at the discretion of the physician. The change from enrollment (at least 1 month after starting treatment with paricalcitol iv) to the 6-month post-enrollment visit was calculated as the 6-month post-enrollment visit value minus the enrollment value.
Time Frame: Enrollment, 6 months
Population: All enrolled participants with available data at the study timepoints, regardless of whether or not they completed the study (i.e., the 6-month post-enrollment follow-up).
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
pg/mL
  Enrollment (n=250) | 423.4 (331.5)
  6 months post-enrollment (n=218) | 390.8 (332.6)
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p = 0.02, Wilcoxon signed rank test-paired samples; Mean Difference (Final Values) = -21.4, Standard Deviation 324.8 — n= 215 (paired samples)

17. Secondary Outcome: Change Per Month From Baseline to 6 Months in Parathyroid Hormone (PTH) Levels (pg/mL Per Month)
Description: PTH levels were recorded at each study visit prior to hemodialysis according to routine clinical practice and at the discretion of the physician. Linear models based on Generalized Estimating Equations (GEE) were used to assess the effect of time on change from enrollment (at least 1 month after starting treatment with paricalcitol iv) through 3 months post-enrollment and 6 months post-enrollment.
Time Frame: Enrollment, 3 months post-enrollment, 6 months post-enrollment
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: pg/mL per month
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Number analyzed (Participants) | 254
pg/mL per month | -5.66 [-12.80 to 1.48]
Statistical Analysis 1: Comparison: Chronic Kidney Disease, Secondary Hyperpathyroidism; Test type: Superiority or Other; p = 0.12, Generalized Estimating Equation approach; Generalized Estimating Equation approach (autoregressive structure)

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from enrollment to 30 days after study completion (7 months).
Description: Of the 265 participants enrolled, 11 participants were considered to have protocol deviations and were excluded from the enrolled population and from all study-related analyses. A total of 254 participants were included in all of the study analyses.
Groups:
- Chronic Kidney Disease, Secondary Hyperpathyroidism: All eligible patients treated with paricalcitol iv according to the approved Summary of Product Characteristics (SmPC)
Arm/Group | Chronic Kidney Disease, Secondary Hyperpathyroidism
Serious Adverse Events (participants affected / at risk) | 28/254
Other Adverse Events (participants affected / at risk) | 0/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Kidney Disease, Secondary Hyperpathyroidism (N=254)
Cardiac arrest (Cardiac disorders) | 12
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Sudden death (Cardiac disorders) | 1
Hematocrit decreased (Investigations) | 3
Blood parathyroid hormone decreased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
Prothrombin time prolonged (Investigations) | 1
Red blood cell sedimentation rate increased (Investigations) | 1
Weight decreased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Pyrexia (General disorders) | 2
Condition aggravated (General disorders) | 1
Death (General disorders) | 1
Fatigue (General disorders) | 1
Inflammation (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Hematochezia (Gastrointestinal disorders) | 1
Large intestinal polyp (Gastrointestinal disorders) | 1
Pancreatic pseudocyst (Gastrointestinal disorders) | 1
Peritoneal hemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Ischemic stroke (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
Peripheral coldness (Vascular disorders) | 1
Peripheral ischemia (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Vasodilatation (Vascular disorders) | 1
Sepsis (Infections and infestations) | 2
Arteriovenous graft site abscess (Infections and infestations) | 1
Bacteremia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 2
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Loss of consciousness (Nervous system disorders) | 2
Coma (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Grand mal convulsion (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Unresponsive to stimuli (Nervous system disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hematuria (Renal and urinary disorders) | 1
Kidney rupture (Renal and urinary disorders) | 1
Arteriovenous graft (Surgical and medical procedures) | 1
Nephrectomy (Surgical and medical procedures) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Ascites (Hepatobiliary disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic encephalopathy (Hepatobiliary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Agitation (Psychiatric disorders) | 1
Communication disorder (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Dry gangrene (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.